CLINICAL TRIAL: NCT05511584
Title: Oxygen Consumption and Sevoflurane Uptake Based on Physiological Dead Space Estimation During Closed Circuit Anesthesia: A Prospective Interventional Study
Brief Title: Oxygen Consumption and Sevoflurane Uptake Based on Physiological Dead Space Estimation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VO2.SEVOup.VDphys
Record Dates: First submitted 2022-08-18; First posted 2022-08-23 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Oxygen Consumption; Sevoflurane; Anesthetics, Inhalation; Surgery
Keywords: Oxygen Consumption; Sevoflurane; Anesthesia, Closed-Circuit
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VO2 and SEVOup (Experimental): Estimation of VO2 and SEVOup (ml/min) followed by estimation of O2 and sevoflurane supply (DO2 and SEVOsuppl, respectively) through a closed-circuit anesthesia administration system.
  Interventions: Procedure: VO2 estimation; Procedure: SEVOup estimation

INTERVENTIONS:
Procedure: VO2 estimation — 1. st) VO2 (ml/min) will be estimated based on the formula: Inspired fraction of O2 (FiO2) - Expired fraction of O2 (FeO2) * minute volume (Volmin)
  2. nd) Assuming the estimation of VDphys obtained with Fluxmed®, the investigators will calculate the VO2 corresponding to effective alveolar ventilation (VO2.alv), which will be the result of subtracting VDphys from Volmin.
  3. rd) The investigators will calculate the O2 delivered fraction (DO2) (ml/min) corresponding to the estimated VO2.alv, and will supply it to the system while working in a closed-circuit mode.
Procedure: SEVOup estimation — 1. st) SEVOup (ml/min) will be estimated based on the formula: Inspired fraction of sevoflurane (Fi.sevo) - Expired fraction of sevoflurane (Fe.sevo) * Volmin
  2. nd) Assuming the estimation of VDphys obtained with Fluxmed®, the investigators will calculate the SEVOup corresponding to effective alveolar ventilation (SEVOup.alv), which will be the result of subtracting VDphys from Volmin.
  3. rd) The investigators will calculate the sevoflurane delivered fraction (SEVOsuppl) (ml/min) corresponding to the estimated SEVOup.alv, and will supply it to the system while working in a closed-circuit mode.

SUMMARY:
In this study, the investigators will evaluate whether the delivered fraction of oxygen (O2) and sevoflurane administered through a a closed circuit and calculated on the basis of the estimations of O2 consumption (VO2) and sevoflurane uptake (SEVOup) through the inspired-expired fraction gradients of both gases once subtracted the physiological dead space (VDphys), adequately fits the real gases consumption. All participants will be ventilated under a tailored open lung approach (tOLA) strategy.

DETAILED DESCRIPTION:
The "quantity" of the lung that participates in gas exchange in anesthetized and mechanically ventilated patients varies depending on individual conditions. This "part" of the lung that is responsible for "breathing" is referred as the respiratory volume in contrast to that "part" or volume of the lung that is in charge of driving the air towards the respiratory zones: the trachea, bronchi, et cetera, which do not directly participate in breathing. This conduction volume, together with that alveolar volume excluded from gas exchange due to different circumstances, constitutes the physiological dead space (VDphys), which represents the percentage of tidal volume that does not participate of respiration. The VDphys can be estimated by different means.

Knowing the VDphys will allow the clinicians to more precisely adjust the amount of oxygen and anesthetic gas (sevoflurane) to be supplied to the anesthesia workstation when working in a closed circuit mode, given that the estimations of VO2 and SEVOup, and consequently of the milliliters of oxygen and sevoflurane to supply per minute (DO2 and SEVOsuppl, respectively), are calculated in the basis of the "respiratory" volume rather that in the "total" tidal volume (TV); this is, taking in consideration the VDphys/TV ratio.

In this work, the investigators will evaluate the accuracy in estimating VO2 and SEVOup taking into consideration the VDphys/TV ratio when working with a closed circuit mode of anesthesia administration. The investigators will study the relationship between the DO2 and SEVOsuppl, calculated based on VDphys/TV ratio, and the real consumption of O2 and sevoflurane measured through the gas analyzer of the anesthesia workstation.

Methods

This one-arm interventional study corresponds to phase 3 of the study "Influence of Inspiratory Pause on Ventilatory Efficiency in Robotic Surgery. A Prospective Paired Study". Participants will be consecutively recruited among those patients submitted to prostatic robotic surgery, once obtained the corresponding informed consent. The study will be carried out in a tertiary care teaching hospital (Hospital Universitario Virgen del Rocío). Approval for this study will be sought from the local ethics committee. The recruitment will be made on investigators availability.

Study protocol Participants will be ventilated through a Primus anesthesia workstation (Drager, Telford, PA, USA) using a TV of 7 mL/kg of predicted body weight. The ventilation mode used will be volume control, which will include an inspiration: expiration ratio of 1:2 and a respiratory rate of 12-15 breaths/min to maintain carbon dioxide (CO2) at the end of expiration (etCO2) between 35 and 40 mmHg and an initial positive end expiratory pressure (PEEP) of 5 cmH2O. A 30 % end inspiratory pause will be scheduled for all participants. A fresh gas flow of 0.5 to 1 L/min with an inspired fraction of oxygen (FIO2) of 0.5 will be used throughout the procedure. Anesthesia will be maintained with remifentanil 0.03 to 0.05 µg/kg/min and sevoflurane, with a minimum alveolar concentration of 0.6 to 0.8, which will be adjusted to the patient's age to ensure a Bispectral Index (BIS Quatro; Covidien Ilc , Mansfield, MA, USA) between 40-60. Rocuronium will be administered to ensure deep neuromuscular blockade during the study, which will be monitored by train of four neuromuscular relaxation (TOF-watch®, Organon Ltd., Swords, Co. Dublin, Ireland). A tOLA strategy will be applied ten minutes after commencing mechanical ventilation, and it will comprise an alveolar recruitment manoeuver (ARM) with titration of optimal PEEP (PEEPop) on a decremental PEEP trial, followed by a new ARM and setting a tailored open-lung PEEP (tOL-PEEP), that 2 cm H2O higher than PEEPop. All ventilation parameters will remain stable throughout the study except PEEP, which will be titrated according to the principles of tOLA.

A Fluxmed® monitor (MBMED, Buenos Aires, Argentina) will be used for volumetric capnography. The data will be downloaded to a laptop after proper calibration of the flow and pressure sensors. The computer, through the FluxView software (MBMED, Buenos Aires, Argentina), will automatically calculate the following parameters:alveolar, airway and physiological dead spaces (VDalv, VDaw and VDphys, respectively) and its values related to the TV. The anesthesia workstation will be used for continuous monitoring of airway pressures and inspired and expired fraction of the gases administered. The investigators will measure VO2 and SEVOup while applying a low flow anesthesia administration method.

Statistical analysis will be performed by the principal investigator. For data analysis, the statistical software IBM SPSS Statistics for Windows, version 24 (IBM Corp., Armonk, NY, USA) will be used. The investigators will perform an exploratory analysis of the data, using the mean ± standard deviation or the median with interquartile range for quantitative variables. The investigators will use percentages for the analysis of qualitative variables and will check the normality of data distribution with the Kolmogorov-Smirnov test or with the Shapiro-Wilk test for variables with less than 50 records. The Student's t test for paired samples will be used to study the behavior of the quantitative variables at different times (intragroup comparisons). The investigators will also study the correlation between the consumption and uptake estimations (VO2 and SEVOup, respectively) measured as milliliters per minute (ml/min), and the ml/min delivered of both gases through the closed-circuit anesthesia system.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (≥ 18 years) scheduled for robotic prostatic surgery at the investigators´ institution
* Written informed consent

Exclusion Criteria:

* Participation in another interventional study
* Participants unable to understand the information contained in the informed consent
* American Society of Anesthesiologists (ASA) classification grade = IV
* Patient in dialysis
* Chronic obstructive pulmonary disease (COPD) grade Global Initiative for Chronic Obstructive Lung Disease(GOLD) > 2
* Functional vital capacity < 60% or > 120% of the predicted
* Body mass index (BMI) > 35 kg/m2
* Relation arterial pressure of oxygen (PaO2)/FiO2 <200 mmHg in the baseline sample
* Presence of mechanical ventilation in the 72 hours prior to enrollment
* New York Heart Association (NYHA) functional class ≥ 3
* Clinically suspected heart failure
* Diagnosis or suspicion of intracranial hypertension
* Presence of pneumothorax or giant bullae on preoperative imaging tests
* Use of Continuous Positive Airway Pressure (CPAP).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in FeO2 during the closed-circuit ventilation mode | Intraoperative ( From the beginning of the maintenance phase of the anesthesia , with recording every 10 minutes or at any time if a deviation of the end-tidal fraction of O2 higher than 5% of the estimated value is detected)
  Any deviation of the expired fractions of O2 (FeO2) with respect to the reference value (this calculated based on VO2.alv estimation). The investigators will reflect this potential deviation through time.
Change in Fe.sevo during the closed-circuit ventilation mode | Intraoperative (From the beginning of the maintenance phase of the anesthesia , with recording every 10 minutes or at any time if a deviation of the end-tidal fraction of sevoflurane higher than 5% of the estimated value is detected)
  Any deviation of the expired fraction of sevoflurane (Fe.sevo) with respect to the reference value (this calculated based on SEVOup.alv estimation). The investigators will reflect this potential deviation through time.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel de la Matta, MD, Principal Investigator — Hospitales Universitarios Virgen del Rocío
Locations (1):
- Hospital Universitario Virgen del Rocío, Seville, Spain